CLINICAL TRIAL: NCT01556945
Title: Phase I/IIa Safety, Immunogenicity, and Preliminary Efficacy of an Administration Schedule of FMP1 and SmithKlineBeecham Biologicals' Candidate Malaria Vaccine RTS,S Each Adjuvanted With SBAS2, Given Concomitantly in Separate Injections
Brief Title: Safety and Preliminary Efficacy of the Malaria Vaccine Candidates Falciparum Merozoite Protein-1 (FMP1) and SmithKlineBeecham (SKBB) Candidate Malaria Vaccine RTS,S
Acronym: MAL019
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: WRAIR #849
Record Dates: First submitted 2012-03-14; First posted 2012-03-19 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-05

CONDITIONS: Malaria, Falciparum
Keywords: P. falciparum; vaccine; healthy volunteers
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group A : FMP1/AS02 + RTS,S/AS02 (Experimental): FMP1 malaria vaccine given with the GlaxoSmithKline (GSK) adjuvant system, number 2 (AS02) and a second experimental malaria vaccine RTS,S also given with AS02 adjuvant concomitantly as separate sites of injection on days 0, 28 and 84. Malaria challenge phase began 14-30 days after the last vaccine.
  Interventions: Biological: FMP1/AS02; Biological: RTS,S/AS02; Other: Malaria challenge
- Group B : FMP1/AS02 + RTS,S/AS02 (Experimental): FMP1 malaria vaccine given with the adjuvant AS02 and a second experimental malaria vaccine RTS,S also given with AS02 adjuvant at one injection site and saline at the opposite site on days 0, 28 and 84. Malaria challenge phase began 14-30 days after the last vaccine.
  Interventions: Biological: FMP1/AS02; Biological: RTS,S/AS02; Other: Malaria challenge
- Group C: FMP1/AS02 + AS02 (Experimental): FMP1 malaria vaccine given with the adjuvant AS02 and a second experimental malaria vaccine RTS,S also given with adjuvant AS02 adjuvant alone at one injection site and saline at the opposite site on days 0, 28 and 84. Malaria challenge phase began 14-30 days after the last vaccine.
  Interventions: Biological: FMP1/AS02; Other: AS02 adjuvant alone; Other: Malaria challenge
- Group D : RTS,S/AS02 + AS02 (Experimental): RTS,S malaria vaccine given with the adjuvant AS02 and an adjuvant AS02 alone concomitantly at separate sites of injection on days 0, 28 and 84. Malaria challenge phase began 14-30 days after the last vaccine.
  Interventions: Biological: RTS,S/AS02; Other: AS02 adjuvant alone; Other: Malaria challenge
- Control cohort (Placebo Comparator): Infectivity controls (unvaccinated). Non-randomized infectivity controls were recruited specifically for the malaria challenge phase of the trial.
  Interventions: Other: Malaria challenge

INTERVENTIONS:
Biological: FMP1/AS02 — The vaccine antigen FMP1 consists of a recombinant histidine-tagged (His6) fusion protein expressed in E. coli. The lyophilized pellet contained per vaccine vial 62.5 μg merozoite surface protein-142 (MSP-142) with 3.1% lactose as cryoprotectant in each 3 ml monodose vial. The pellet was reconstituted with AS02.
  Arms: Group A : FMP1/AS02 + RTS,S/AS02; Group B : FMP1/AS02 + RTS,S/AS02; Group C: FMP1/AS02 + AS02
Biological: RTS,S/AS02 — The vaccine antigen RTS,S, is a recombinant subunit vaccine produced in, and purified from yeast cells. The final lyophilized pellet contained 62.5 μg RTS,S with 3.15% lactose as cryoprotectant per 3 ml monodose vial. The pellet was reconstituted in AS02 and each 0.5 ml dose contained 50 μg RTS,S.
  Arms: Group A : FMP1/AS02 + RTS,S/AS02; Group B : FMP1/AS02 + RTS,S/AS02; Group D : RTS,S/AS02 + AS02
Other: AS02 adjuvant alone — AS02 adjuvant contains 50 μg monophosphoryl lipid A (MPL) and 50 μg Quillaja saponaria 21 (QS-21), 250 μl of SB62 (oil/water emulsion) in phosphate buffered saline (PBS) per volume of 0.5 ml.
  Arms: Group C: FMP1/AS02 + AS02; Group D : RTS,S/AS02 + AS02
Other: Malaria challenge — Experimental challenge homologous strain of P.falciparum sporozoites. Mosquitoes infected with malaria approximately 17 to 19 days earlier and that contained sporozoites in their salivary glands. For each volunteer, five mosquitoes were allowed to feed over five minutes, after which they were dissected to confirm how many were infected, and the salivary glands scored.

SUMMARY:
The purpose of this study is to see if two new malaria vaccines called FMP1 and RTSS, combined with an adjuvant (called SBAS2) which helps stimulate the body's immune system, are safe, demonstrate an immune response through blood tests, and lastly, to see if the vaccines can prevent malaria infection.

The RTS,S vaccine contains a malaria protein in combination with a portion of the commercially available hepatitis B vaccine. The FMP1 vaccine also contains a malaria protein. The adjuvant called SBAS2, is a special oil in water emulsion. Vaccinations are done at study days 0, 28 and 84, followed by a malaria challenge approximately 14 days after the 3rd vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult, 18-45
* Available for duration of study (9 months)
* Written informed consent prior to any study procedures

Exclusion Criteria:

* Prior receipt of an investigational malaria vaccine or one containing MPL or QS-21
* Use of any investigational or non-registered drug/vaccine or planned administration of vaccine not foreseen by study protocol; each issue within 30 days preceding the first dose of study vaccine
* Administration of chronic immunosuppressants
* Chronic use of antibiotics
* History of malaria ever, or use of malaria chemoprophylaxis within 60 days prior to vaccination
* Known exposure to malaria within the past 12 months or planned travel to malarious area during the study period
* Confirmed or suspected immunosuppressive or immunodeficient condition
* Family history of congenital or hereditary immunodeficiency
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine
* Chronic or active neurologic disease including seizures
* History of splenectomy
* Seropositive for hepatitis B or hepatitis C or Human Immunodeficiency Virus (HIV), or other abnormal labs such as significant anemia, elevated creatinine
* Hepatomegaly, or right upper quadrant abdominal pain
* Pregnant or lactating female
* Chronic or active drug or alcohol use
* History of severe reactions to mosquito bites
* Any history of anaphylaxis to vaccinations

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2001-04; Primary Completion 2002-02 (Actual)

PRIMARY OUTCOMES:
Safety | two years
  Measured through adverse event collection and immunogenicity results

CONTACTS AND LOCATIONS:
Locations (1):
- WRAIR Clinical Trials Center, Silver Spring, Maryland, United States

REFERENCES:
- [Derived] Cummings JF, Polhemus ME, Kester KE, Ockenhouse CF, Gasser RA Jr, Coyne P, Wortmann G, Nielsen RK, Schaecher K, Holland CA, Krzych U, Tornieporth N, Soisson LA, Angov E, Heppner DG; RTS,S Vaccine Evaluation Group. A phase IIa, randomized, double-blind, safety, immunogenicity and efficacy trial of Plasmodium falciparum vaccine antigens merozoite surface protein 1 and RTS,S formulated with AS02 adjuvant in healthy, malaria-naive adults. Vaccine. 2024 Apr 30;42(12):3066-3074. doi: 10.1016/j.vaccine.2024.03.072. Epub 2024 Apr 6. PMID 38584058